CLINICAL TRIAL: NCT03659045
Title: Double-blind, Randomized, Multicenter Study Evaluating 200 Mg Versus 600 Mg of Mifegyne® on Pain in Medical Termination of Pregnancy (MToP) Up to 7 Weeks of Amenorreha (WA). DoMy Study.
Brief Title: Pain Assessment in MToP Up to 7 WA (during 5h After Misoprostol Intake)
Acronym: DoMy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-53
Record Dates: First submitted 2018-08-17; First posted 2018-09-06 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2023-07

CONDITIONS: Abortion-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mifegyne® 600MG (Experimental): Patients assigned to this group will receive three 200 mg tablets of Mifegyne® taken during the consultation Patients will answer to a scale of pain
  Interventions: Other: scale of pain
- Mifegyne® 200MG (Placebo Comparator): Patients assigned to this group will receive one 200 mg Mifegyne® tablet and two placebo tablets that will be taken during the consultation.
  Patients will answer to a scale of pain
  Interventions: Other: scale of pain

INTERVENTIONS:
Other: scale of pain — The measurement is simple, reproducible, performed using a scale of pain rated from 0 to 10 (0 absence of pain, 10 maximum of pain felt)

SUMMARY:
In 2016, medical termination of pregnancy represent 64% of total abortions in France. Thus, it is a frequent act involving a large majority of women and a health-care public subject. The two medicines used in medical abortion are mifepristone and misoprostol. The efficacy of mifepristone-misoprostol combination is very high, greater than 90% up to 7 SA. Medical abortion may be performed in outpatient basis or in short-terme hospitalization. One of the limits of this technique development is the pain caused by the drugs intake mainly due to the uterine contractions induced by misoprostol intake. Thus it is recommended a systematic analgesics intake but despite these guidelines, pain level reported by the patients remains significant. There is very limited data on the misoprostol influence or mifepristone dose on pain. In a recent observational multicenter study, mifepristone 600 mg was reported to be associated with decreased pain compared with mifepristone 200 mg.

In this context, it is important to confirm by a higher level evidence of study that the protocol using mifepristone 600 mg decreases the pain level of medical abortion compared to a protocol using mifepristone 200 mg. In the absence of benefit, we will not be able to conclude to a benefit on the prevention of pain with a protocol associating 600 mg of mifepristone and 400 μg of misoprostol. If the benefit on pain is confirmed, it will be interesting to evaluate the efficacy / pain ratio of the 200 mg and 600 mg dose in terms of quality of care or medical and economic impact.

The clinical study is interventional, prospective, comparative, randomized, double-blind, multi-center, conducted in 11 French hospitals carrying out voluntary medical termination of pregnancy.

The data will be collected by the physician during the 4 consultations (initial consultation of abortion request, inclusion consultation with Mifegyne® intake, consultation of misoprostol intake (short-terme hospitalization), follow-up consultation from the available data in the patient's medical file and from the questionning and clinical examination data made during these 4 consultations.

DETAILED DESCRIPTION:
Background and purpose of the study: In 2015, the voluntary interruption of medication pregnancy represented 57% of the total number of abortions in metropolitan France, ie 116,000 annual acts. Thus, it is a frequent act involving a very large majority of women and a subject of public health. The two molecules used in drug-induced abortion are mifepristone and misoprostol. The efficacy of mifepristone-misoprostol combination is very high, greater than 90% before 7 SA. One of the limits of the diffusion of this technique is the pain caused by the drug intake mainly at the time of the uterine contractions induced by the taking of misoprostol. Thus it is recommended a systematic taking of analgesics but despite these recommendations the level of pain reported by the patients remains high. There is very little data on the influence of the dose of misoprotol or mifepristone on pain. In a recent multicenter observational study, mifepristone 600 mg was reported to be associated with a decrease in pain compared with 200 mg while the misoprostol dose had no influence.

In this context, it is important to confirm by a higher level of evidence study whether the protocol using 600 mg mifepristone decreases the pain level of drug-induced abortion compared to a protocol using 200 mg, at the same dose of misoprostol .

MATERIAL AND METHODS: A prospective, randomized, double-blind, multi-center clinical study, conducted in metropolitan France, in 11 hospital centers performing drug-induced abortion involving 320 patients. The inclusion criteria will be patients requesting a drug-induced abortion, agreeing to participate in the study and not having a contraindication to both study drugs. The main criterion will be the pain felt within 5 hours after taking misoprostol. The secondary criteria will be the pain felt and painkillers consumed during the various stages of drug induced abortion, the failure rate, the number of intermediate consultations, tolerance and quality of life.

Expected results and consequences: In the absence of benefit, the investigators will not be able to conclude to a benefit on the prevention of the pain with a protocol associating 600 mg of mifepristone and 400 μg of misoprostol. In the event of confirmation of benefit on pain, it will be interesting to evaluate the efficacy / pain ratio of the 200 mg and 600 mg dose in terms of the quality of care or the medical and economic impact.

ELIGIBILITY:
Inclusion Criteria:

* Woman aged 18 or over.
* A woman with a single intrauterine pregnancy, whose term is less than 7 weeks on the day of taking mifegyne, estimated by ultrasound with a measurement of the craniocaudal length less than or equal to 10 millimeters.
* Woman wishing a drug induced abortion in hospital.
* Woman having signed a written informed consent and pledging to respect the instructions of the protocol.

Exclusion Criteria:

* Minor woman.
* Women with multiple pregnancy, uterine malformation (septate uterus, cocked hat, fibroids) or a coagulation disorder defined by biological parameters (TP <70%, TCA patient / control ratio <1.20).
* Women with a contraindication to mifepristone: chronic adrenal insufficiency, severe asthma not controlled by treatment, hereditary porphyria, known allergy to the active substance or to any of the excipients.
* Women with a contraindication to misoprostol: hypersensitivity to the active substance, to any of the excipients or to other prostaglandins;
* Women presenting a contraindication to one of the analgesics used in the study (nefopam, paracetamol, opium, caffeine).
* Woman with suspected ectopic pregnancy
* Woman with pregnancy not confirmed by ultrasound or biology
* Woman with a contraindication to the antiemetic potentially used (ondansetron)
* Women with a contraindication to lactose
* Patients undergoing treatment with one or more CYP3A4-moderate or potent drugs
* Female not affiliated to the social security scheme.
* Women having not signed informed consent.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — aborption
Enrollment: 320 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2023-03-22 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Pain assessment in MToP up to 7 WA after Mifegyne® intake | During 5 hour after Mifegyne® intake
  Pain measurement is simple, reproducible, performed by numeric scale rated from 0 to 100 (0 no pain, 100 maximum pain felt). The scale will be explained to the patient

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO PRADALIE, Study Director — APHM
Locations (8):
- France (8):
  - Assistance Publique Des Hopitaux de Marseille, Marseille, PACA
  - Chu Grenoble Alpes, Grenoble
  - Hospices Civils de Lyon, Lyon
  - Centre Hospitalier Du Belvedere, Mont-Saint-Aignan
  - Centre Clotilde Vautier de L'Union de Gestion de La Clinique Jules Verne de Nantes, Nantes
  - Assistance Publique Hôpitaux de Paris, Paris
  - Centre Hospitalier de Roubaix, Roubaix
  - Chu de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No